CLINICAL TRIAL: NCT01608607
Title: Effect of Fructose-containing Sugar Sweetened Beverages (SSBs) on Body Weight: A Systematic Review and Meta-analysis of Controlled Feeding Trials to Provide Evidence-based Guidance for Nutrition Guidelines Development
Brief Title: Meta-analysis of Fructose-Containing Sugar Sweetened Beverages (SSBs) and Weight Change
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: John Sievenpiper (Other)
Collaborators: Calorie Control Council (Other); Canada Research Chairs Endowment of the Federal Government of Canada (Other Government); Canadian Institutes of Health Research (CIHR) (Other Government)
Responsible Party: Sponsor-Investigator, John Sievenpiper, Adjunct Research Fellow, University of Toronto
Organization: University of Toronto (Other)
Other Study IDs: CCC 2012 KRS
Record Dates: First submitted 2012-05-14; First posted 2012-05-31 (Estimated); Last update posted 2015-05-27 (Estimated); Status verified 2015-05

CONDITIONS: Overweight; Obesity; Diabetes; Prediabetes; Dysglycemia; Metabolic Syndrome
Keywords: Systematic review and meta-analysis; Evidence-based medicine (EBM); Evidence-based nutrition (EBN); Clinical practice guidelines; Clinical trials; Dietary sugars; Fructose; High fructose corn syrup; sucrose; Isocaloric; Hypercaloric; Glycemic control; Insulin resistance; Body weight; body mass index; waist circumference
MeSH Terms: conditions — Overweight; Obesity; Diabetes Mellitus; Prediabetic State; Metabolic Syndrome; Insulin Resistance; Body Weight

STUDY DESIGN:
Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Other: Fructose-containing sugar sweetened beverages — Oral dietary fructose-containing sugar sweetened beverages in isocaloric exchange for other sources of carbohydrate (isocaloric trials) or hypercaloric exchange for beverages containing a non-nutritive sweetener or added to a control diet as a source of excess energy (hypercaloric trials)

SUMMARY:
Since uncontrolled observational studies first linked fructose to the epidemic of obesity almost a decade ago, it has become a focus of intense concern regarding its role in the obesity epidemic. Despite the uncertainties in the evidence,the recommendations of international health organizations have cautioned against moderate to high intakes fructose-containing sugars, especially those from sugar sweetened beverages (SSBs). To improve the evidence on which nutrition recommendations are based, the investigators propose to study of the effect of fructose-containing sugar sweetened beverages (SSBs)on body weight, by undertaking a systematic synthesis of the data taken from all available clinical studies in humans. This technique has the strength of allowing all of the available data to be pooled together and differences to be explored in groups of different study participants (healthy humans of different sex, weight, and age and in those with diseases which predispose to disturbances in metabolism, such as diabetes) with dietary fructose in different forms, doses, and with differing durations of exposure. The findings generated by this proposed knowledge synthesis will help improve the health of consumers through informing recommendations for the general public, as well as those at risk of diabetes and cardiovascular disease.

DETAILED DESCRIPTION:
Background: Fructose has become a focus of intense concern regarding its links to the obesity epidemic. There have been dozens of editorials, commentaries, and letters in the scientific literature and numerous pieces in the lay and social media calling for efforts to restrict its intake and even regulate it like tobacco or alcohol. Uncontrolled observational studies which have linked increasing fructose intake with increasing obesity rates since the 1970s and animal models of fructose overfeeding at levels of exposure far beyond actual population levels of intake have been used to underpin this debate. Evidence from observational studies and controlled feeding trials also suggest a positive association between the consumption of fructose-containing sugar-sweetened beverages, in which high fructose corn syrup (HFCS) is the main sweetener, and increased energy consumption and weight gain, but not all meta-analyses have supported this conclusion. Despite the limitations in extrapolating from these data and their inconsistency with data from controlled trials in humans (the highest level of evidence used in evidence based medicine), the American Heart Association (AHA) have taken a risk reduction approach to added fructose-containing sugars, especially those from sugar sweetened beverages (SSBs), setting highly restrictive upper thresholds for their intake to achieve and maintain healthy body-weights.

Objective: To improve the evidence on which recommendations and public health policy are based, we propose to conduct a systematic review and meta-analysis of the effect of fructose-containing SSBs on body weight in controlled feeding trials.

Design: The planning and conduct of the proposed meta-analyses will follow the Cochrane handbook for systematic reviews of interventions. The reporting will follow the Preferred Reporting Items for Systematic reviews and Meta-Analyses (PRISMA) guidelines.

Data sources. MEDLINE, EMBASE, CINAHL and The Cochrane Central Register of Controlled Trials (Clinical Trials; CENTRAL) will be searched using appropriate search terms, supplemented by manual, hand searches of bibliographies.

Study selection: We will include controlled feeding trials investigating the effect of fructose-containing (fructose, sucrose, and HFCS) SSBs in isocaloric exchange for other carbohydrate sources (isocaloric trials) or hypercaloric exchange for beverages containing a non-nutritive sweetener or added to a control diet as a source of excess energy (hypercaloric trials) on body weight in humans. Studies that are <7-days diet duration, lack a control, or do not provide viable endpoint data will be excluded.

Data extraction. Two investigators will independently extract information about study design, sample size, subject characteristics, fructose form, dose, reference-carbohydrate, follow-up, and background diet profile. Mean±SEM values will be extracted for body weight. Standard computations and imputations will be used to derive missing variance data. The quality/validity of each study will be assessed using the Heyland Methodological Quality Score (MQS).

Ouctomes: Body weight change will be the only ouctome.

Data synthesis. Meta-analyses will be conducted using the Generic Inverse Variance method applying random effects models expressed as standardized mean differences (SMDs) with 95% CIs. Paired analyses will be applied for crossover trials. Heterogeneity will be assessed by the Q statistic and quantified by I2. Sensitivity analyses and a priori subgroup analyses will be undertaken to explore sources of heterogeneity including the effect of underlying disease status, sugar type (fructose, sucrose, HFCS), reference carbohydrate (comparator), fructose form, dose, follow-up, study design, baseline measurements, and study quality on the effect of fructose. Significant unexplained heterogeneity will be investigated by additional post hoc subgroup analyses (e.g. age, sex, level of feeding control, energy balance and composition of the background diet, etc.). Meta-regression analyses will assess the significance of subgroups analyses. Publication bias will be investigated by inspection of funnel plots.

Knowledge translation plan: The results will be disseminated through interactive presentations at local, national, and international scientific meetings and publication in high impact factor journals. Target audiences will include the public health and scientific communities with interest in nutrition, diabetes, obesity, and cardiovascular disease. Feedback will be incorporated and used to improve the public health message and key areas for future research will be defined. Applicant/Co-applicant Decision Makers will network among opinion leaders to increase awareness and participate directly as committee members in the development of future guidelines.

Preliminary findings: We conducted a systematic review and meta-analysis to investigate the effect of dietary fructose on body weight in controlled feeding trials (Sievenpiper et al. Ann Intern Med. 2012;156:291-304). We identified 31 isocaloric trials (n=635), in which fructose was exchanged for the same amount of carbohydrate in the diet, and 10 hypercaloric trials (n=119), in which the diet was supplemented with excess energy from high-dose fructose. Whereas there was no effect of fructose under isocaloric trial conditions, fructose under hypercaloric trial conditions (+104-250-g/day, +18-97% energy) significantly and consistently increased weight (MD=0.53-kg or 1.17-lb [95%CI: 0.26 to 0.79-kg or 0.57 to 1.74-lb]). In both analyses, fructose behaved no differently than sucrose or HFCS, where these sugars were the comparators, and fructose in fluid (beverage) form did not increase body weight in the isocaloric trials. We concluded that the available trials did not support a body weight raising-effect of fructose in isocaloric exchange for other carbohydrate. There was, however, consistent evidence for a modest body weight raising-effect of fructose at extreme doses providing excess energy, where the effect of energy appeared to be dominant. The implications of our findings for "real world" dietary advice was complicated by the fact that sucrose and HFCS are the primary fructose-containing sweeteners in the US diet. The proposed systematic review and meta-analysis will address this limitation directly by investigating the effect of all fructose-containing (fructose, sucrose, and HFCS) SSBs.

Significance: The proposed project will aid in knowledge translation related to the effects of dietary fructose on overweight and obesity, strengthening the evidence-base for recommendations and improving health outcomes through informing consumers and guiding future research.

ELIGIBILITY:
Inclusion Criteria:

* Trials in humans
* Oral fructose intervention
* Suitable control (i.e. another carbohydrate source in isocaloric exchange for fructose or a control diet which is compared with the same diet supplemented with excess energy from fructose)
* >= 7-days diet duration
* Viable endpoint data

Exclusion Criteria:

* Non-human studies
* IV or parenteral fructose
* High fructose corn syrup or sucrose intervention (except where these are the comparators)
* Lack of a suitable control
* < 7-days diet duration.
* No viable endpoint data

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Varied
Sampling Method: Probability Sample
Enrollment: 1 (Actual)
Dates: Start 2012-05; Primary Completion 2014-09 (Actual); Study Completion 2015-10 (Estimated)

PRIMARY OUTCOMES:
Body weight | 1.5-years

CONTACTS AND LOCATIONS:
Overall Officials: John L Sievenpiper, MD, PhD, Study Director — Department of Pathology and Molecular Medicine, McMaster University and Clinical Nutrition and Risk Factor Modification Centre, St. Michael's Hospital; Russell J de Souza, ScD, RD, Study Director — Department of Epidemiology and Biostatistics, McMaster University and Clinical Nutrition and Risk Factor Modification Centre, St. Michael's Hospital; David JA Jenkins, MD, PhD, DSc, Principal Investigator — Department of Nutritional Sciences and Medicine, University of Toronto and Clinical Nutrition and Risk Factor Modification Centre, St. Michael's Hospital
Locations (1):
- The Toronto 3D (Diet, Digestive tract and Disease) Knowledge Synthesis and Clinical Trials Unit, Clinical Nutrition and Risk Factor Modification Centre, St. Micheal's Hospital, Toronto, Ontario, Canada

REFERENCES:
- [Background] Sievenpiper JL, de Souza RJ, Mirrahimi A, Yu ME, Carleton AJ, Beyene J, Chiavaroli L, Di Buono M, Jenkins AL, Leiter LA, Wolever TM, Kendall CW, Jenkins DJ. Effect of fructose on body weight in controlled feeding trials: a systematic review and meta-analysis. Ann Intern Med. 2012 Feb 21;156(4):291-304. doi: 10.7326/0003-4819-156-4-201202210-00007. PMID 22351714
- [Background] Sievenpiper JL, Chiavaroli L, de Souza RJ, Mirrahimi A, Cozma AI, Ha V, Wang DD, Yu ME, Carleton AJ, Beyene J, Di Buono M, Jenkins AL, Leiter LA, Wolever TM, Kendall CW, Jenkins DJ. 'Catalytic' doses of fructose may benefit glycaemic control without harming cardiometabolic risk factors: a small meta-analysis of randomised controlled feeding trials. Br J Nutr. 2012 Aug;108(3):418-23. doi: 10.1017/S000711451200013X. Epub 2012 Feb 21. PMID 22354959
- [Background] Ha V, Sievenpiper JL, de Souza RJ, Chiavaroli L, Wang DD, Cozma AI, Mirrahimi A, Yu ME, Carleton AJ, Dibuono M, Jenkins AL, Leiter LA, Wolever TM, Beyene J, Kendall CW, Jenkins DJ. Effect of fructose on blood pressure: a systematic review and meta-analysis of controlled feeding trials. Hypertension. 2012 Apr;59(4):787-95. doi: 10.1161/HYPERTENSIONAHA.111.182311. Epub 2012 Feb 13. PMID 22331380
- [Background] Wang DD, Sievenpiper JL, de Souza RJ, Chiavaroli L, Ha V, Cozma AI, Mirrahimi A, Yu ME, Carleton AJ, Di Buono M, Jenkins AL, Leiter LA, Wolever TM, Beyene J, Kendall CW, Jenkins DJ. The effects of fructose intake on serum uric acid vary among controlled dietary trials. J Nutr. 2012 May;142(5):916-23. doi: 10.3945/jn.111.151951. Epub 2012 Mar 28. PMID 22457397
- [Background] Sievenpiper JL, de Souza RJ, Jenkins DJ. Sugar: fruit fructose is still healthy. Nature. 2012 Feb 22;482(7386):470. doi: 10.1038/482470e. No abstract available. PMID 22358823
- [Background] Sievenpiper JL, de Souza RJ, Kendall CW, Jenkins DJ. Is fructose a story of mice but not men? J Am Diet Assoc. 2011 Feb;111(2):219-20; author reply 220-2. doi: 10.1016/j.jada.2010.12.001. No abstract available. PMID 21272692
- [Background] Sievenpiper JL, Carleton AJ, Chatha S, Jiang HY, de Souza RJ, Beyene J, Kendall CW, Jenkins DJ. Heterogeneous effects of fructose on blood lipids in individuals with type 2 diabetes: systematic review and meta-analysis of experimental trials in humans. Diabetes Care. 2009 Oct;32(10):1930-7. doi: 10.2337/dc09-0619. Epub 2009 Jul 10. PMID 19592634